CLINICAL TRIAL: NCT05171829
Title: An Educational Self-tracking Tool for Identification of SARS-CoV-2 Risk Transmission: a Randomised Controlled Trial
Brief Title: An Educational Self-tracking Tool for Identification of SARS-CoV-2 Risk Transmission
Acronym: TrackU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Escoles Universitaries Gimbernat (Other); University of Barcelona (Other); Barcelona Institute for Global Health (Other); Universitat Politècnica de Catalunya (Other); Universitat Oberta de Catalunya (Other)
Responsible Party: Principal Investigator, Anna Llupia, Public Health Specialist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCB/2021/1054
Record Dates: First submitted 2021-12-21; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Sars-CoV-2 Infection; Empowerment; Transmission
MeSH Terms: conditions — COVID-19; Empowerment

STUDY DESIGN:
Masking Description: Statistician masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention : Educational tool (Experimental): self-tracking educational tool (diary)
  Interventions: Other: Track U
- Control (No Intervention)

INTERVENTIONS:
Other: Track U — Track U diary
  Arms: Intervention : Educational tool

SUMMARY:
One way to empower a community, in epidemic control issues, is to know the first-hand screening tools. There are no evaluations of these home-use tools from the perspective of patient and citizen empowerment and participation. The main objective of this study is to analyze whether a self-tracking and self-tracing tool, developed in a participatory way, increases the risk identification of the disease and the empowerment in terms of risk management of transmission by the participants.

ELIGIBILITY:
Inclusion Criteria:

Fluent in Catalan or Spanish, Resident in Catalonia, Signs informed consent, Commitment to use the tool if he/she gets in intervention group.

Exclusion Criteria:

Language barrier and other conditions that do not allow self-completion of the survey Be a COVID case or contact at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-12-27 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Risk identification of SARS-CoV 2 transmission | 17 days
  Risk identification of SARS-CoV 2 transmission

SECONDARY OUTCOMES:
Empowerment in SARS-CoV 2 transmission | 17 days
  Empowerment in SARS-CoV 2 transmission

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided